CLINICAL TRIAL: NCT00543413
Title: A Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Study to Assess the Efficacy and Tolerability of MK8141 in Hypertensive Patients
Brief Title: A Study to Determine the Effectiveness and Tolerability of MK8141 in Patients With High Blood Pressure (MK-8141-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8141-006; MK8141-006; 2007_587
Record Dates: First submitted 2007-10-05; First posted 2007-10-15 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — MK-8141; Enalapril; Enalaprilat

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental): Arm 1: Drug 250 mg
  Interventions: Drug: MK8141
- 2 (Experimental): Arm 2: Drug 500 mg
  Interventions: Drug: MK8141
- 3 (Active Comparator): Arm 3: Active Comparator
  Interventions: Drug: Enalapril
- 4 (Placebo Comparator): Arm 4: Pbo Comparator
  Interventions: Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: MK8141 — MK8141 250 mg tablet once daily; 500 mg tablet once daily 4 week treatment period
  Arms: 1; 2
Drug: Comparator: placebo (unspecified) — MK8141 Pbo tablet once daily. 4 week treatment period.
  Arms: 4
Drug: Enalapril — Enalapril 20 mg tablet once daily. 4 week treatment period.
  Other Names: Vasotec®
  Arms: 3

SUMMARY:
This study will evaluate the effectiveness and tolerability of MK8141 in lowering blood pressure in patients who have hypertension (high blood pressure).

ELIGIBILITY:
Inclusion Criteria:

* You are 35 to 65 years of age
* In the past 14 days you have not been treated for hypertension
* In the past 14 days you have not taken more than 2 medications to treat high blood pressure
* You are a woman who is not able to have children or do not use birth control

Exclusion Criteria:

* You are taking more than 2 medications to treat high blood pressure
* You have a history of a stroke, transient ischemic attack (TIA), heart attack, congestive heart failure, coronary artery bypass surgery
* You have Type 1 or 2 diabetes mellitus
* You have an active liver disease, gallbladder disease, or bowel disease
* You are HIV positive
* You have certain types of cancer
* You abuse drug or alcohol
* You have participated in another clinical study in last 4 weeks

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To measure the tolerability and effectiveness of MK8141 in lowering 24-hour mean ambulatory blood pressure versus placebo after 4 weeks of treatment. | after 4 weeks of treatment

SECONDARY OUTCOMES:
Compare MK8141 versus placebo in lowering 24-hour mean sitting blood pressure by ambulatory blood pressure monitoring and in lowering trough mean sitting diastolic and systolic blood pressure after 4 weeks of treatment. | after 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Jones-Burton C, Rubino J, Roy S, Mai Y, Meehan A, Bellet M, Feig P. Effects of the renin inhibitor MK-8141 (ACT-077825) in patients with hypertension. J Am Soc Hypertens. 2010 Sep-Oct;4(5):219-26. doi: 10.1016/j.jash.2010.06.006. Epub 2010 Aug 12. PMID 20705534